CLINICAL TRIAL: NCT06326138
Title: Pharmacokinetics and Pharmacodynamics of Edoxaban in Subjects With Severe Obesity Before and After Sleeve Gastrectomy and Roux-en-Y Gastric Bypass
Brief Title: Pharmacokinetics and Pharmacodynamics of Edoxaban Before and After Bariatric Surgery
Acronym: EXPOSE
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No support form the sponsor
Sponsor: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Paul Poirier, MD, PhD, Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22121
Record Dates: First submitted 2024-03-11; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Intervention Model Description: Group 1: 12 patients waiting for a sleeve gastrectomy surgery and 12 patients waiting for a Roux-en-Y gastric bypass surgery.
  Group 2: 12 patients 12 months after Roux-en-Y gastric bypass surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Roux en Y gastric bypass and Sleeve Gastrectomy (Experimental): Edoxaban pharmacodynamic and pharmacokinetic will be evaluated before and 48 ± 5 hours after bariatric surgery (sleeve gastrectomy and Roux-en-Y gastric bypass).
  Interventions: Drug: Edoxaban Pharmacokinetics and Pharmacodynamics
- Group 2 - Roux en Y gastric bypass (Experimental): Edoxaban pharmacodynamic and pharmacokinetic will be evaluated at 12 ± 3 months following Roux-en-Y gastric bypass surgery.
  Interventions: Drug: Edoxaban Pharmacokinetics and Pharmacodynamics

INTERVENTIONS:
Drug: Edoxaban Pharmacokinetics and Pharmacodynamics — Participants will be received single oral doses of edoxaban 60 mg.

SUMMARY:
The study will be conducted at a single site in the Canada, Quebec. Participants will be recruited from the bariatric surgery clinic and will be required to be either, waiting for sleeve gastrectomy surgery (n=12, restrictive bariatric surgery, Group 1) or Roux-en-Y gastric bypass (n=12, mixed bariatric surgery, Group 1), or had underwent Roux-en-Y gastric bypass 12 ± 3 months ago (n=12, Group 2).

Participants in Group 1, edoxaban pharmacokinetic and pharmacodynamics will be evaluated before and 48 ± 5 hours after bariatric surgery (sleeve gastrectomy and Roux-en-Y gastric bypass). Participants in Group 2, edoxaban pharmacokinetic and pharmacodynamics will be evaluated only once, at 12 ± 3 months following their Roux-en-Y gastric bypass.

All participants will be received single oral doses of 60 mg edoxaban at each pharmacokinetic and pharmacodynamics evaluation.

DETAILED DESCRIPTION:
Screening visit (Group 1 and 2: visit 1) // Group 1: Screening will take place within 3 to 4-months window before bariatric surgery. Group 2: Screening will take place within 1-months window approximately 12± 3 months after bariatric surgery.

Informed consent will be obtained from the subject prior to performing any of the screening assessments.

The following activities and/or assessments will be performed at/during Screening: Informed consent, Inclusion/exclusion criteria, Medical history, Concomitant medications, Physical examination, including height, weight, and body mass index (BMI), Blood and urine samples, 12-lead ECG, Vital signs.

Pharmacokinetic (PK) and pharmacodynamics (PD) visit Group 1: PK and PD visit will take place after the screening visit and within 3-months window before bariatric surgery as well as 48 hours after bariatric surgery.

Group 2: PK and PD visit will take place after the screening visit and within 1-months window after bariatric surgery (12± 3 months).

On PK and PD visit, the following procedures will be performed: Vital signs, ECG, Concomitant medications, Edoxaban dosing (before 8:00 AM), Pharmacokinetics (PK) and Pharmacodynamics (PD) blood draws (predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours), Post dose fasting and water restrictions, as appropriate, Adverse event (AE) monitoring.

Follow-up 1 - Group 1 and Group 2: Follow-up 1 will take place onsite 24 hours after PK and PD visits.

On follow-up 1, the following procedures will be performed: PK and PD blood draws, Concomitant medications, AE monitoring.

Follow-up 2 - Group 1 and Group 2: Follow-up 2 will be a phone contact and will take place 7 days after PK and PD visits.

On follow-up 2, the following procedures will be performed: Concomitant medications, AE monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects over 18 years of age.
2. Females who are of non-childbearing potential must be:

   * Surgically sterile (i.e., bilateral tubal ligation or removal of both ovaries and/or uterus at least 6 months prior to dosing).
   * Naturally postmenopausal (spontaneous cessation of menses) for at least 12 consecutive months prior to screening visit, with a follicle stimulating hormone level in the postmenopausal range.
3. Females of childbearing potential must have a negative urine pregnancy test at each study visit with PK and PD evaluation.
4. Subjects must agree not to donate blood, plasma, platelets, or any other blood components for 4 weeks before each study visit with PK and PD evaluation.
5. Subjects must agree to food and drug restrictions during the study.
6. Subjects must agree to abstain from alcohol, cola, tea, coffee, chocolate, and other caffeinated drink and food from 2 days before each study visit with PK and PD evaluation.
7. Subjects must agree to abstain from food and beverages containing grapefruit, grapefruit juice, cranberry juice, lime, pomelo, marmalade and Seville oranges from 10 days before each study visit with PK and PD evaluation.
8. Absence of clinically significant deviations from medical history, physical examination and 12-lead ECG, as deemed by the Investigator, prior to enrollment.
9. Subject must have sinus rhythm on the 12-lead ECG at each study visit with PK and PD evaluation.
10. Has given written informed consent prior to participating in the study.
11. Able to understand and willing to comply with all study requirements, and willing to allow the collection of all blood specimens.
12. Normal coagulation values from INR (< 1.2).

Exclusion Criteria:

1. History or current evidence of clinically significant cardiac, hepatic, renal, pulmonary, endocrine, neurologic, infectious, gastrointestinal, hematologic, or oncologic disease as determined by screening medical history, physical examination, or 12-lead ECG.
2. Subjects with QTcF interval duration > 450 msec for males and >470 for females.
3. Subjects with abnormal waveform morphology on any of the ECGs at the screening that would preclude accurate measurement of the QT interval duration.
4. Subjects with a resting systolic (treated) blood pressure > 159 mmHg or < 90 mmHg or a diastolic blood pressure > 95 mmHg or < 50 mmHg.
5. History of malignancy.
6. Subjects who have had a clinically significant illness within 4 weeks prior to the first dose.
7. Subjects who have used any drugs or substances known to be strong inhibitors or strong inducers of CYP 3A4/5 enzymes or P-gp within 28 days prior to the first dosing.
8. Subjects with history of major bleeding, major trauma, or major surgical procedure of any type within 6 months of dosing.
9. Subjects with history of peptic ulcer, gastrointestinal bleeding (including hematemesis, melena, rectal bleeding) or bleeding from hemorrhoids.
10. Subjects with history of thrombophlebitis or pulmonary embolism.
11. Subjects with history of minor bleeding episodes such as epistaxis, rectal bleeding (spots of blood on toilet paper), and gingival bleeding within 3 months before the first dose.
12. Subjects who have any family history (suspected or documented) of coagulopathy.
13. Females with a history of dysfunctional uterine bleeding, including history of menorrhagia (heavy menstrual bleeding), metrorrhagia, or polymenorrhea.
14. Subjects with eye surgeries or trauma to the head or eye within 14 days of the first dose.
15. Subjects who have used fish oil, acetylsalicylic acid, any over-the-counter medication containing acetylsalicylic acid, nonsteroidal anti-inflammatory drugs (NSAIDs), or other supplements (e.g., gingko biloba, …) that could prolong bleeding within 14 days of the first dose or expect to use these during the study.
16. Subjects who have used anticoagulants (i.e., warfarin, low molecular weight heparin [LMWH]), coagulants, anti-platelet (i.e., clopidogrel) 30 days prior to the first dose.
17. Subjects with abnormal complete blood count at screening.
18. Subjects with estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2.
19. Subject is currently enrolled in or has not yet completed at least 30 days or 5 half-lives, whichever is longer, since ending another investigational device or drug study or is receiving other investigational agents.
20. Subjects who, in the opinion of the Investigator, should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics edoxaban parameter | 0 hour (before taking edoxaban) - 0.5 hours - 1 hour - 1.5 hours - 2 hours - 2.5 hours - 3 hours - 4 hours - 6 hours - 8 hours - 12 hours - and 24 hours after taking edoxaban
  Maximum edoxaban plasma concentration
Pharmacokinetics edoxaban parameter | 0 hour (before taking edoxaban) - 0.5 hours - 1 hour - 1.5 hours - 2 hours - 2.5 hours - 3 hours - 4 hours - 6 hours - 8 hours - 12 hours - and 24 hours after taking edoxaban
  Time to reach maximum edoxaban plasma concentration
Pharmacokinetics edoxaban parameter | 0 hour (before taking edoxaban) - 0.5 hours - 1 hour - 1.5 hours - 2 hours - 2.5 hours - 3 hours - 4 hours - 6 hours - 8 hours - 12 hours - and 24 hours after taking edoxaban
  Area under the edoxaban plasma concentration-time curve
Pharmacokinetics edoxaban parameter | 0 hour (before taking edoxaban) - 0.5 hours - 1 hour - 1.5 hours - 2 hours - 2.5 hours - 3 hours - 4 hours - 6 hours - 8 hours - 12 hours - and 24 hours after taking edoxaban
  Edoxaban half time

SECONDARY OUTCOMES:
Pharmacodynamics edoxaban parameter | 0 hour (before taking edoxaban) - 0.5 hours - 1 hour - 1.5 hours - 2 hours - 2.5 hours - 3 hours - 4 hours - 6 hours - 8 hours - 12 hours - and 24 hours after taking edoxaban
  aPTT
Pharmacodynamics edoxaban parameter | 0 hour (before taking edoxaban) - 0.5 hours - 1 hour - 1.5 hours - 2 hours - 2.5 hours - 3 hours - 4 hours - 6 hours - 8 hours - 12 hours - and 24 hours after taking edoxaban
  PT/INR
Pharmacodynamics edoxaban parameter | 0 hour (before taking edoxaban) - 0.5 hours - 1 hour - 1.5 hours - 2 hours - 2.5 hours - 3 hours - 4 hours - 6 hours - 8 hours - 12 hours - and 24 hours after taking edoxaban
  anti-FXa activity

CONTACTS AND LOCATIONS:
Overall Officials: Paul Poirier, MD, Phd, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval

IPD SHARING:
Plan to Share IPD: No